CLINICAL TRIAL: NCT03364517
Title: Evaluation of a Standardized Medical Regulation Strategy on the Reduction of Deliveries Outside Medical Presence.
Brief Title: Extra Hospital Delivery Outside Medical Presence.
Acronym: REGUL-AIpM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital NOVO (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CHRD1616
Record Dates: First submitted 2017-11-23; First posted 2017-12-06 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2022-08

CONDITIONS: Delivery
Keywords: Medical regulation; SPIA; Imminent delivery

STUDY DESIGN:
Intervention Model Description: Randomized controlled cluster study.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group SPIA (Experimental): The regulator will be asked to systematically use the tool Predictor score of the imminence of a childbirth (SPIA). This tool is used to evaluate the means to be sent following a call for imminent delivery outside the hospital.
  Interventions: Other: Predictor score of the imminence of a childbirth (SPIA)
- Control group (No Intervention): The classic care will be made according to the usual practices of the doctor and the center.

INTERVENTIONS:
Other: Predictor score of the imminence of a childbirth (SPIA) — The SPIA score is based on the analysis of 6 types of criteria: panic during the call, the possibility of having a telephone contact with the parturient, the urge to push and if so for how long, the rhythm of the CU, some aggravating factors (history of fast delivery or at home, maternal age between 26 and 35 years, lack of follow-up of pregnancy) and 2 minor factors (nulliparity and the taking of a tocolytic treatment). Each criteria is between 0 to 8, except for the 2 minor criteria for which 7 and 3 points are removed if they are present. This gives a score between -10 and +33, which is weighted according to the admission time estimated at the hospital (30 minutes, 1h and 2h).
  Arms: Experimental group SPIA

SUMMARY:
The purpose of this study is to prospectively evaluate a standardized procedure of medical regulation based on a validated predictive score of eminent delivery (SPIA) in comparison with usual inhomogeneous practices. This standardized procedure impacting the process of care production (when receiving the call for regulation for unannounced delivery) would improve the quality of care of parturients while rationalizing the use of medical teams in the field.

DETAILED DESCRIPTION:
This study aims to evaluate a standardized procedure of medical regulation based on a validated predictive score of eminent delivery (SPIA) in comparison with usual inhomogeneous practices. It will therefore focus on the issues of medical regulation at SAMU - Center 15. The goal of the regulator is to provide the right care in situations of constrained medical resources, that is to say the need to bring the right answer in the most appropriate time and to direct the parturient in the structure which is the most adapted. Currently, very few studies are conducted in this area. However, maternal and fetal morbidity out off medical presence exists and deserves special attention. Unexpected childbirth outside a maternity ward is an emergency for the mother and the child, with maternal-fetal excess mortality 2 to 3 times higher. In this area, the modalities of response to the call - after assessment by the regulator of the foreseeable delay of delivery - are very unequal in France. The hypothesis of this study is that a decision-making aid using score SPIA will provide better management by reducing the risk of delivery without the presence of a doctor or midwife.

The expected benefits for the patients are a decrease in the maternal-fetal morbidity and mortality, an adapted orientation of the patient according to the foreseeable delay before delivery. This is to avoid the patient's referral to a maternity ward that is not her own when it is not necessary - that is, an orientation in a maternity ward that is inappropriate for her condition and / or with a risk of delivery outside maternity. Finally, another expected benefit is the patient delivery in the presence of a doctor and / or midwife.

The expected benefits for public health are an adapted sending of means, principle of the "just care" and the good use of the medical resources, to avoid the situations of deficiency of SMUR following an inappropriate sending (accessibility of the offer of care) and improved practices, without additional cost to public health (improve the efficiency of the UAS regulation - Center 15).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman over 33 WA
* Age ≥ 18 years
* Calling the regulation of SAMU-Center 15 for start of work
* Patient not planning to give birth at home
* Delivery not having started at the time of the first call (hair, head, buttocks or feet not visible)
* Absence of a doctor, obstetrician or midwife on the spot during the call
* French language included (Patient and / or Near)

Exclusion Criteria:

* Opposition of the patient after sending the information note.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8208 (Actual)
Dates: Start 2018-03-14 (Actual); Primary Completion 2021-12-14 (Actual); Study Completion 2021-12-14 (Actual)

PRIMARY OUTCOMES:
Number of deliveries without the presence of a doctor or midwife and absence of the SMUR sent in first intention. | Through study completion, an average of eighteen months.
  It will be the number of unexpected deliveries out of medical presence.

SECONDARY OUTCOMES:
Number of deliveries outside maternity. | Through study completion, an average of eighteen months.
  This is the number of deliveries that took place outside the maternity ward. For the included participants, the investigators divide the number of deliveries that took place outside the maternity ward by the number of births that took place in the maternity ward. It is then sufficient to multiply the result by one hundred to obtain the percentage that the investigators wish to measure.
Number of adapted responses. | Through study completion, an average of eighteen months.
  It is the number of patients who have obtained a response adapted to their condition, that is to say the provision of resources corresponding to the recommendations in relation to the expected delay until delivery.
Duration of the call collected on the regulation. | At the moment of inclusion of the patient, an average one day.
  The investigators measure the duration in minutes of the call collected on the regulation file before sending the appropriate means to the state of the participant. This is the time in minutes between the time the investigator takes the call and the time the decision is made.
Regulatory investigator satisfaction by a standardized questionnaire. | Through study completion, an average of six months.
  This consists of measuring the satisfaction of the investigator by a standardized questionnaire for the study. This questionnaire contains only one question: what is the difficulty you had in making the regulatory decision? Then just check the corresponding box. These boxes are ten in number. The zero box corresponds to no difficulty in making the decision and box 10 corresponds to the maximum difficulty in making the decision.
APGAR scores of newborn at birth and 10 minutes of delivery. | At one minute then at ten minutes.
  The APGAR score is used to assess the condition of a newborn. It is measured once at birth and a second time ten minutes after delivery. The optimal state of the baby gives a score equal to ten. The apparent state of death is zero side. It allows investigators to determine the course of action and the surveillance elements of each newborn. A score between seven and ten consists of a conduct of the investigators that will be mild and will consist of a simple unclogging of the airways and an optional oxygen supply. A score between four and seven will consist of serious care that is needed and in the absence of rapid improvement the child will be unblocked, receive oxygen in the mask and be infused. Finally, a score lower than four will lead to intensive resuscitation maneuvers that will be undertaken and in the absence of dramatic improvement the child will be transferred to a resuscitation unit.
Vital status of mother and newborn (at 3 days). | Three days after delivery.
  This is to collect the vital status of the mother and newborn three days after delivery.
Number of hypothermia, hypoglycemia, respiratory and circulatory distress, hospitalizations in intensive care-neonatology, among newborns. | An average of one month after delivery.
  The investigators collect the number of newborns who have experienced episodes of hypothermia, hypoglycemia, respiratory and circulatory distress and hospitalizations in intensive care-neonatology.

CONTACTS AND LOCATIONS:
Overall Officials: Agnès RICARD-HIBON, Principal Investigator — Hôpital NOVO
Locations (19):
- France (19):
  - Centre Hospitalier René-DUBOS, Cergy-Pontoise, Cergy-pontoise
  - Centre Hospitalier Universitaire d'Amiens, Amiens
  - Centre Hospitalier Régional Universitaire de Besançon, Besançon
  - Centre Hospitalier Universitaire Avicenne, Bobigny
  - Hôpital Pellegrin, Bordeau
  - Centre Hospitalier Henri Mondor, Créteil
  - Centre Hospitalier Universitaire de Dijon, Dijon
  - Centre Hospitalier Universitaire de Grenoble, Grenoble
  - Hôpital André Mignot, Le Chesnay
  - Centre Hospitalier Régional Universitaire de Lille, Lille
  - Groupement Hospitalier Edouard Herriot, Lyon
  - Centre Hospitalier Marc Jacquet, Melun
  - Centre Hospitalier Régional Mets-Thionville, Metz
  - Centre Hospitalier Annecy-Genevois, Metz-Tessy
  - Centre Hospitalier Universitaire de Nancy, Nancy
  - Centre Hospitalier Universitaire de Rennes, Rennes
  - Centre Hospitalier Universitaire de la Réunion, Saint-Denis
  - Centre Hospitalier de Toulon, Toulon
  - Hôpital Purpan, Toulouse

IPD SHARING:
Plan to Share IPD: No